CLINICAL TRIAL: NCT04445740
Title: Feasibility, Acceptability, and Preliminary Efficacy of the i Heart Rhythm Project
Brief Title: The i Heart Rhythm Project: Healthy Sleep and Behavioral Rhythms for Obesity Prevention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Jennette P. Moreno, Assistant Professor, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: H-47369; R00HD091396 (NIH)
Record Dates: First submitted 2020-05-26; First posted 2020-06-24 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Obesity Prevention

STUDY DESIGN:
Who Masked: Investigator
Masking Description: key personnel will be masked
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants will receive an intervention and will participate in assessments
  Interventions: Behavioral: i♥rhythm project
- Control (No Intervention): Participants will not receive an intervention, but will participate in assessments

INTERVENTIONS:
Behavioral: i♥rhythm project — behavioral mobile health intervention, targeting parents of 5-8 year olds, designed to promote consistent behavioral rhythms in children through consistent bedtimes, light exposure, meal timing, and physical activity.
  Arms: Intervention

SUMMARY:
This pilot study will examine the feasibility, acceptability, and preliminary efficacy of the intervention. This will ensure that all aspects of the research protocol and procedures work as desired and are acceptable to families in preparation for the fully powered randomized controlled trial. The proposed study will assess our ability to: 1)recruit, consent, and retain participants, 2) deliver the intervention, 3) implement study and assessment procedures 4) assess the reliability of the proposed measures in this sample, 5) determine whether modifications to the intervention, procedures, and measures are needed prior to conducting a fully powered study, and 6) willingness of participants to participate in the intervention.

DETAILED DESCRIPTION:
The current study employs a 2 group randomized control design (treatment and no-treatment control) with randomization occurring after baseline (time 0) and 3 additional evaluation periods (end of intervention (time 1), and 9 months (time 2) and 12 months post intervention (time 3)). Because the the i♥rhythm project is intended to prevent children from beginning a trajectory toward overweight/obesity in elementary school, the impact of the intervention on change in standardized BMI (BMIz) during the following summer (time 2 and 3) will be explored, identifying whether a maintenance intervention is needed. Following the intervention and final data assessment (time 1 and 3), qualitative interviews will explore the acceptability of the intervention, treatment barriers and facilitators, difficulties with study procedures, maintenance of improvements, and self-efficacy to maintain improvements. A third treatment condition controlling for the effect of attention was beyond the scope of the current feasibility study.

ELIGIBILITY:
Inclusion Criteria:

* The index child is 5-8 years old and currently enrolled in kindergarten, first, or second grade
* Parent reports being a daily user of social media
* Parent willing to engage in an mobile health intervention that includes social media
* Parent owns a smart phone
* At least 1 parent is comfortable participating in the intervention and responding to questionnaires in English
* Index child has a BMI >50th percentile
* families live in the greater Houston area and able to attend in-person data collection at the Children's Nutrition Research Center.

Exclusion Criteria:

* Per parent report, the child does not have a chronic medical condition affecting sleep, eating behaviors, weight status, or behavioral rhythms (e.g., obstructive sleep apnea, attention deficit hyperactivity disorder, autism). The inclusion and exclusion criteria will be assessed using a screening questionnaire and assessments which will be administered following the consenting procedures.
* Per parent report, the child is not being treated with a medication or supplement known to affect sleep.
* Child has not participated in an obesity prevention or obesity treatment program in the last 6 months
* Child had not been retaine 2 or more grades for academic reason or has intellectual difficulities that would influence their ability to complet questionnaires or participate in interviews.

Ages: 5 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 92 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2023-08-18 (Actual); Study Completion 2023-08-18 (Actual)

PRIMARY OUTCOMES:
Feasibility Criteria: ability to recruit the needed sample size | 3 months
  The feasibility of the intervention will be established by our ability to recruit the needed sample size and retain at least 80% at Time 1 and 60% at Time 3; favorable acceptability ratings by 80% of the sample, participation in greater than 60% of daily diaries, views of intervention materials by 80% of participants. Decisions regarding changes to the intervention will be made based on the attainment of feasibility criteria and post-assessment interviews. Decisions regarding changes to the intervention will be made based on the attainment of feasibility criteria and post-assessment interviews.
Treatment Acceptability | 3 months
  Treatment Acceptability Report Form-Revised(TARF-R) 185 is a 20-item global measure of treatment acceptability for behavioral interventions. The TARF-R has demonstrated good internal consistency (αs>.69) and evidence of construct validity. A favorable rating is considered 4 or greater.

SECONDARY OUTCOMES:
Anthropometrics | 0 months, 3 months, 12 months and 15 months
  Body Mass Index (BMI) is the most common indicator of body size and has been consistently correlated with metabolic problems in children. Participants' height and weight will be measured using established protocols. BMI (kg/m2) will be computed and BMI %ile and BMIz will be calculated from age and gender normative data. BMI %ile will determine weight status group. Change in BMI and BMIz are the best proxy measures for change in fat mass and standardized fat mass and will assess exploratory hypotheses. Change in BMI will serve as the primary outcome for the fully powered randomized controlled trial. For the current application, feasibility criteria will serve as the primary outcome.
Measurement of endogenous circadian rhythms | 0 months, 3 months, 12 months and 15 months
  Circadian phase can be examined by measuring the circadian timing of melatonin onset under dim light conditions (dim light melatonin onset; DLMO). Compared to markers of endogenous circadian rhythms, melatonin is relatively robust. Salivary DLMO measures have demonstrated high intraclass correlations (.93) with plasma and sensitivity and specificity comparable to plasma assays. Following established procedures with children, salivary DLMO will be collected on a weekday evening in the laboratory under dim light conditions (<40 lux), via a cheek swab every hour beginning 5 hours prior to and ending 1 hour following typical bedtime. Saliva samples will be centrifuged, frozen, and assayed using radioimmunoassay test kits. DLMO phase will be determined using linear interpolation across the time points before and after melatonin concentration increased to and remained above 4pg/mL.
Actigraphy for the measurement of sleep, sleep/wake patterns, physical activity, and light exposure. | 0 months, 3 months, 12 months and 15 months
  Actigraphs (GT3X-BT, Pensacola, FL) worn on the wrist of the dominant hand 24 hours a day for 7 days will measure sleep duration and timing of sleep onset and waking. Wrist placement reliably measures sleep duration in adolescents. Sleep diaries will be completed. Monitor-wear logs will identify times the accelerometer is removed and the activity engaged in while the monitor is off. The photocell contained in the Actigraph GT3X-BT will be used to measure ambient light exposure. Accelerometers have been extensively used to assess children's physical activity (PA). Five days of monitoring had 0.8 reliability of accurately capturing the habitual PA of children. Activity counts captured in 5-second epochs will be categorized into sedentary, light, moderate, and vigorous PA using established cut points.
Body composition | 0 months, 3 months, 12 months and 15 months
  Since BMI can misrepresent adiposity among muscular and slender children, use of additional body fat indicators has been recommended. Investigators will assess percent body fat using Bod Pod.
Dietary Assessment | 0 months, 3 months, 12 months and 15 months
  The Automated Self-Administered 24-Hour Dietary Assessment Tool (ASA-24)174 will be used to assess children's dietary intake (e.g., total daily caloric intake, timing of intake, timing of the last eating episode of the day). As recommended, parents will complete the adult version of the ASA-24, providing proxy report of their child's dietary intake. Investigators will use 3 days of diet assessment as 3 days optimize the prediction of doubly labeled water estimated energy expenditure.
Parenting Structure | 0 months, 3 months, 12 months and 15 months
  Comprehensive General Parenting Questionnaire (CGPQ) is a parent report of parenting practices among parents of 5-13 year olds. Investigators will assess subscales related to parenting structure (inconsistent discipline, consistency, organization, and scaffolding). There is support for the construct validity of the CGPQ. Parenting structure subscales have demonstrated acceptable to good internal reliability (ranging from .67-.74). Subscale scores range from 5 to 25. Higher scores indicate higher levels of structure.
Bedtime Routines | 0 months, 3 months, 12 months and 15 months
  The Bedtimes Routines Questionnaire (BRQ), is a 31-item parent report measure of children's bedtime routines, comprised of three scales measuring consistency of bedtime routines (weekday & weekend), reactivity to changes in bedtime routines, and frequency of adaptive and maladaptive activities. The BRQ scales had good internal consistency ranging from α = 0.69 to 0.90. Scores on the consistency and adaptive behavior subscales range from 10 to 50 with higher scores reflecting more consistent bedtime routines and higher. The reactivity scale scores range from 5 to 25 with higher scores reflecting greater reactivity. The maladaptive behavior scale has possible scores ranging from 6 to 30 with higher scores reflecting more maladaptive behaviors.
Summer Care Arrangements | 0 months, 3 months, 12 months and 15 months
  How Children Spend their Summer (e.g., children's involvement in summer school, child care, entertainment programs, as well as day or overnight camps) will be assessed by a parent report survey based on a modified version of the Early Childhood Longitudinal Program Kindergarten Class' parent interview on summer activities. The Girl's Health Enrichment Multisite Studies demographic protocol will be employed with parents.
Stress (Parent) | 0 months, 3 months, 12 months and 15 months
  Perceived Stress Scale (PSS-10) is a 10-item self-report measure of perceived stress with established acceptable psychometric properties(α's >.70, test-retest criterion coefficient >.7, validated factor structure and evidence of convergent validity). Scores range from 0 to 40 with higher scores reflecting higher levels of perceived stress.
Social Support (Parent) | 0 months, 3 months, 12 months and 15 months
  Interpersonal Support Evaluation List (ISEL) is a 12-item self-report measure of the perceived availability of social support (i.e. Tangible, appraisal, and belonging). The ISEL has demonstrated good reliability. The "tangible" subscale assesses perceived availability of resources and material aid; the "appraisal" subscale assesses the perceived availability of another individual(s) to discuss one's problems; the "self-esteem" subscale assesses the perceived availability of someone to compare one's self to in a positive manner; and the "belonging" subscale, the perceived availability of having others to socialize and do things with. Scores range from 0-30 on each scale with greater scores indicating higher levels of social support.
Motivation to Continue in the Program | 3 months
  The Treatment Questionnaire Concerning Continued Program Participation was originally developed to assess reasons for continuing to participate in a weight-loss program. We have adapted it assess reasons for continuing to participate focused on addressing children's sleep during summer. Scores in the Autonomous Regulation scale range from 5 to 35 and scores on the Controlled Regulation range from 8 to 56. Higher scores reflect higher levels of Autonomous and Controlled regulation.

CONTACTS AND LOCATIONS:
Overall Officials: Jennette Moreno, Principal Investigator — Baylor College of Medicine; Hafza Dadabhoy, MS, Study Director — Baylor College of Medicine
Locations (1):
- Children's Nutrition Research Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moreno JP, Dadabhoy H, Musaad S, Baranowski T, Thompson D, Alfano CA, Crowley SJ. Evaluation of a Circadian Rhythm and Sleep-Focused Mobile Health Intervention for the Prevention of Accelerated Summer Weight Gain Among Elementary School-Age Children: Protocol for a Randomized Controlled Feasibility Study. JMIR Res Protoc. 2022 May 16;11(5):e37002. doi: 10.2196/37002. PMID 35576573
- [Background] Moreno JP, Hannay KM, Walch O, Dadabhoy H, Christian J, Puyau M, El-Mubasher A, Bacha F, Grant SR, Park RJ, Cheng P. Estimating circadian phase in elementary school children: leveraging advances in physiologically informed models of circadian entrainment and wearable devices. Sleep. 2022 Jun 13;45(6):zsac061. doi: 10.1093/sleep/zsac061. PMID 35275213